CLINICAL TRIAL: NCT05318040
Title: Phase 1 Study Evaluating Safety and Tolerability of Escalating Single and Multiple Doses of CMS121 and Food Effect in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of CMS121, a Drug Candidate for Alzheimer's Disease, in Healthy Subjects
Acronym: CMS121
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virogenics, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: VG-CMS121-101; R01AG074447 (NIH)
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a 4-Part study. Parts 1, 2, and 3 are randomized, double blind, placebo-controlled investigations of SAD (Part 1) and MAD (Part 2) in healthy young adult subjects and multiple doses in healthy elderly subjects (Part 3) of orally administered CMS121. Part 4 is an open label, 2 way crossover study to assess the effect of food on a single oral dose of CMS121 in healthy young adult subjects.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Single ascending dose - CMS121 (Experimental): Subjects will receive a single oral dose of CMS121 under fed conditions.
  Interventions: Drug: CMS121
- Single ascending dose - placebo (Placebo Comparator): Subjects will receive a single oral dose of placebo under fed conditions.
  Interventions: Drug: Placebo
- Multiple ascending dose - CMS121 (Experimental): Subjects will receive multiple oral doses of CMS121 once daily (QD) for 7 days under fed conditions.
  Interventions: Drug: CMS121
- Multiple ascending dose - placebo (Placebo Comparator): Subjects will receive multiple oral doses of placebo once daily (QD) for 7 days under fed conditions.
  Interventions: Drug: Placebo
- Multiple ascending dose - Elderly cohort - CMS121 (Experimental): Subjects will receive multiple oral doses of CMS121 once daily (QD) for 7 days under fed conditions.
  Interventions: Drug: CMS121
- Multiple ascending dose - Elderly cohort - placebo (Placebo Comparator): Subjects will receive multiple oral doses of placebo once daily (QD) for 7 days under fed conditions.
  Interventions: Drug: Placebo
- Food Effect - CMS121 (Experimental): On Day 1 of each of 2 treatment periods, a single oral dose of CMS121 will be administered following either a standard high fat/high calorie meal (Treatment A) or an overnight fast (Treatment B), as per each subject's assigned randomization sequence (AB or BA). There will be a washout of at least 7 days between doses.
  Interventions: Drug: CMS121

INTERVENTIONS:
Drug: CMS121 — CMS121 is a small molecule to be delivered orally in capsule form and is a therapeutic drug candidate for treatment of Alzheimer's Disease
  Arms: Food Effect - CMS121; Multiple ascending dose - CMS121; Multiple ascending dose - Elderly cohort - CMS121; Single ascending dose - CMS121
Drug: Placebo — Placebo will be provided as visually matching placebo capsules.
  Arms: Multiple ascending dose - Elderly cohort - placebo; Multiple ascending dose - placebo; Single ascending dose - placebo

SUMMARY:
This is a randomized, double-blind study of CMS121 or placebo given as single and multiple escalating doses in normal healthy subjects. The study will be conducted in 4 parts: Part 1 will be a SAD study enrolling approximately 48 young subjects for a total duration of 36 days. Part 2 will be a MAD study enrolling approximately 32 young subjects for a total duration of 43 days, and Part 3 will be a MAD study enrolling approximately 8 elderly subjects for 43 days. Part 4 will be an open-label SAD cross-over cohort of approximately 12 young subjects in a fed or fasted state to evaluate the effect of food on the bioavailability of CMS121, for a duration of 36 days.

DETAILED DESCRIPTION:
This is a randomized, double-blind study of CMS121 or placebo given as single and multiple escalating doses in normal healthy subjects. The study will be conducted in 4 parts: Part 1 will be a SAD study enrolling approximately 48 young subjects for a total duration of approximately 36 days. Part 2 will be a MAD study enrolling approximately 32 young subjects for a total duration of approximately 43 days, and Part 3 will be a MAD study enrolling approximately 8 elderly subjects for a total duration of approximately 43 days. Part 4 will be an open-label SAD cross-over cohort of approximately 12 young subjects in fed and fasted states to evaluate the effect of food on the bioavailability of CMS121, for a duration of 36 days. Safety will be assessed by periodic measurement of vital signs, physical examinations, electrocardiograms (ECGs), blood and urine lab analyses and occurrence of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

To qualify for enrollment, subjects must meet all of the following inclusion criteria:

All Subjects:

* Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent; willing and able to comply with the study schedule, requirements, and restrictions.
* Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dosing.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at the screening visit.
* In good general health, free from clinically significant medical or psychiatric illness, based on medical/surgical history, physical examination, and clinical laboratory tests.
* All laboratory parameters (serum chemistry, hematology, coagulation, and urinalysis) are within the reference range or considered not clinically significant by the PI, at the screening visit.
* Negative results for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), and Hepatitis C virus (HCV) tests (as outlined in protocol) at the screening visit.
* Female subjects must have negative results for pregnancy test at the screening visit and the first check-in and must not be lactating.
* Able to swallow multiple capsules.
* Adequate venous access in the left or right arm to allow collection of the required blood samples.

Parts 1 (SAD) and 2 (MAD):

* Healthy, adult, male or female, 19-60 years of age, inclusive, at the screening visit.

  * Females of childbearing potential .
  * Females of non-childbearing potential are defined as follows:

    * Individuals who have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

      * hysteroscopic sterilization;
      * bilateral tubal ligation or bilateral salpingectomy;
      * hysterectomy;
      * bilateral oophorectomy. or
    * Individuals who are postmenopausal (PMP) with amenorrhea for at least 1 year prior to the first dosing and follicle stimulating hormone (FSH) serum levels consistent with PMP status.
* Females of childbearing potential and male subjects must follow protocol-specified contraception guidance.
* Vital signs must be within the protocol-specified ranges.
* No presence of a clinically significant ECG abnormality as judged by the PI or qualified designee and as per protocol-specified ranges.

Part 3 (Elderly):

* Healthy, adult, male or female, 65-85 years of age, inclusive, at the screening visit.

  * Females of childbearing potential.
  * Females of non-childbearing potential are defined as follows:

    * Individuals who have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

      * hysteroscopic sterilization;
      * bilateral tubal ligation or bilateral salpingectomy;
      * hysterectomy;
      * bilateral oophorectomy. or
    * Individuals who are postmenopausal (PMP) with amenorrhea for at least 1 year prior to the first dosing and follicle stimulating hormone (FSH) serum levels consistent with PMP status.

or

* Individuals who are PMP with amenorrhea for at least 1 year prior to the first dosing and FSH serum levels consistent with PMP status.

  * Females of childbearing potential and male subjects must follow protocol specified contraception guidance.
  * Vital signs must be within the protocol-specified ranges.
  * QTcF interval is ≤450 msec (males) or ≤470 msec (females) and has ECG findings considered normal or not clinically significant by the PI or designee at the screening visit and prior to the first dosing.

Part 4 (Food Effect):

* Healthy, adult, male or female, 19-60 years of age, inclusive, at the screening visit.

  * Females of childbearing potential.
  * Females of non-childbearing potential are defined as follows:

    * Individuals who have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

      * hysteroscopic sterilization;
      * bilateral tubal ligation or bilateral salpingectomy;
      * hysterectomy;
      * bilateral oophorectomy. or
    * Individuals who are PMP with amenorrhea for at least 1 year prior to the first dosing and FSH serum levels consistent with PMP status.
* Females of childbearing potential and male subjects must follow protocol specified contraception guidance.
* Vital signs must be within the protocol-specified ranges.
* QTcF interval is ≤450 msec (males) or ≤470 msec (females) and has ECG findings considered normal or not clinically significant by the PI or designee at the screening visit and prior to the first dosing.
* Able to completely consume a standardized high-fat/high-calorie breakfast as required by the study protocol.

Exclusion Criteria:

* Subjects who meet any of the following criteria must be excluded from the study:

All Subjects:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of malignancy within the past 2 years, with the exception of adequately treated localized skin cancer (basal cell or squamous cell carcinoma) or carcinoma in-situ of the cervix.
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study in the opinion of the PI or designee.
* Evidence of clinically relevant medical illness including cardiovascular, hematological, psychiatric, gastrointestinal, hepatic, renal, rheumatologic, autoimmune, endocrine, pulmonary, neurologic or dermatologic disorder in the opinion of the PI or designee.
* History of skin rash(es) associated with the use of any medication(s).
* Any condition (e.g., chronic diarrhea) or prior surgery (e.g., gastric bypass) that could interfere with drug absorption, distribution, metabolism, or excretion.
* Clinically significant surgical procedure within 90 days prior to the screening visit.
* Clinically significant acute illness or infection within 14 days prior to the first dosing.
* History of significant drug allergies including a history of anaphylactic reaction.
* Family history of sudden death in an otherwise healthy individual.
* Positive urine cotinine at the screening visit or at first check-in.
* Excessive use of alcohol, defined as weekly intake in excess of 14 units of alcohol (1 unit = 12 fluid ounces of beer, 5 fluid ounces of wine, or 1.5 fluid ounces [1 shot] of distilled spirits or liquor), within 6 months prior to the screening visit.
* Positive test result for alcohol or drugs of abuse at the screening visit or first check-in, or history of alcohol and/or drug abuse within the past 2 years prior to the screening visit.
* Heavy caffeine drinker (defined as consumption of >5 servings of caffeinated beverages [e.g., coffee, tea, cola, energy drinks] per day).
* Refusal to refrain from strenuous physical activity from screening until first check-in.
* Unwillingness to avoid sun and/or phototherapy exposure for 72 hours after the last dose of study drug.
* Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing.
* Use of any investigational drug or device within 30 days or biologics for 90 days (or 5 half-lives of the drug, whichever is the longer) prior to the first dosing, or currently participating in another study of an investigational drug or biologics, or a medical device.
* Loss or donation of >500 mL blood within 56 days prior to study drug administration, or donation of plasma within 30 days prior to the first dosing.
* Employee or family member of the PI, study site personnel, or Sponsor.
* Any other reason that, in the opinion of the PI, would render the subject unsuitable for study enrollment.

Parts 1 (SAD):

* History or presence of:

  * risk factors for Torsade de Pointes (e.g., heart failure, cardiomyopathy, or family history of Long QT Syndrome or sudden unexpected cardiac death at a young age);
  * sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or conduction abnormalities;
  * ischemic heart disease, symptomatic arrhythmias, or poorly controlled hypertension.
  * conditions predisposing to QT prolongation including pathological Q-wave.
* Unable to refrain from or anticipates the use of:

  * any drugs, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing;
  * any drugs known to be significant inducers of CYP enzymes and/or P gp, including St. John's Wort, for 28 days prior to the first dosing. Appropriate sources (e.g., Flockhart Table™) will be consulted to confirm lack of PK/pharmacodynamic (PD) interaction with study drug;
  * any drugs that prolong the QT/QTc interval within 14 days (or 5 half-lives, whichever is longer) prior to the first dosing.
* Allergy to band aids, adhesive dressing, or medical tape.
* Glomerular filtration rate (GFR) ≤ 80 mL/min/1.73 m2, as estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

Part 2 (MAD):

* History or presence of:

  * risk factors for Torsade de Pointes (e.g., heart failure, cardiomyopathy, or family history of Long QT Syndrome or sudden unexpected cardiac death at a young age);
  * sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or conduction abnormalities;
  * ischemic heart disease, symptomatic arrhythmias, or poorly controlled hypertension.
  * conditions predisposing to QT prolongation including pathological Q-wave.
* Unable to refrain from or anticipates the use of:

  * any drugs, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing;
  * any drugs known to be significant inducers of CYP enzymes and/or P gp, including St. John's Wort, for 28 days prior to the first dosing. Appropriate sources (e.g., Flockhart Table™) will be consulted to confirm lack of PK/PD interaction with study drug;
  * any drugs that prolong the QT/QTc interval within 14 days (or 5 half-lives, whichever is longer) prior to the first dosing.
* Is at risk of suicide. Has attempted suicide in the past 12 months or Is at risk of suicide, as determined by the PI, psychiatric interview and/or the baseline C-SSRS.
* Allergy to band aids, adhesive dressing, or medical tape.
* GFR ≤ 80 mL/min/1.73 m2, as estimated by the CKD-EPI equation.

Part 3 (Elderly):

* Is at risk of suicide. Has attempted suicide in the past 12 months or Is at risk of suicide, as determined by the PI, psychiatric interview and/or the baseline C-SSRS.
* Unable to refrain from or anticipates the use of:

  * any drugs, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing. Thyroid hormone replacement medication (refer to protocol) will be allowed;
  * any drugs known to be significant inducers of CYP enzymes and/or P gp, including St. John's Wort, for 28 days prior to the first dosing. Appropriate sources (e.g., Flockhart Table™) will be consulted to confirm lack of PK/PD interaction with study drug.
* GFR ≤ 70 mL/min/1.73 m2, as estimated by the CKD-EPI equation.

Part 4 (Food Effect):

* Is lactose intolerant.
* Unable to refrain from or anticipates the use of:

  * any drugs, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing;
  * any drugs known to be significant inducers of CYP enzymes and/or P gp, including St. John's Wort, for 28 days prior to the first dosing. Appropriate sources (e.g., Flockhart Table™) will be consulted to confirm lack of PK/PD interaction with study drug.
* GFR ≤ 80 mL/min/1.73 m2, as estimated by the CKD-EPI equation.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
Safety: Treatment-emergent adverse events (TEAEs) | From baseline through day 8 for SAD cohorts and through day 15 for MAD cohorts
  Number of participants with TEAEs

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Blood concentration levels of CMS121 | From baseline on day 1 through day 4 for SAD cohorts and through day 10 for MAD cohorts
Pharmacokinetics (PK): Urine concentration levels of CMS121 | From baseline on day 1 through day 4 for SAD cohorts and through day 10 for MAD cohorts.
Safety: Effect on electrocardiographic parameters | From baseline on day 1 and for 24hr post day 1 dose for SAD cohorts; from baseline on day 1 and for 24hr post-dose after day 7 dose for MAD cohorts.
  CMS121 concentration and effect on interval change in QTc (dQTc) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT05318040/ICF_000.pdf